CLINICAL TRIAL: NCT04086602
Title: A Phase 1, Randomised, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Dose Study to Determine the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Food Effect of IZD334 in Healthy Adult Participants as Well as an Open-label Cohort to Confirm the Safety, Pharmacokinetics, and Pharmacodynamics in Adult Patients With Cryopyrin-Associated Periodic Syndromes
Brief Title: Safety and Tolerability, Pharmacokinetic and Pharmacodynamic Study With IZD334
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Inflazome UK Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IZD334-001
Record Dates: First submitted 2019-09-09; First posted 2019-09-11 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Healthy Volunteers; Cryopyrin Associated Periodic Syndrome
MeSH Terms: conditions — Cryopyrin-Associated Periodic Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Healthy volunteer section is double blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single Ascending Dose (Experimental): Once daily oral IZD334 or Placebo
  Interventions: Drug: IZD334; Drug: Placebos
- Multiple Ascending Dose (Experimental): Once or twice daily oral IZD334 or Placebo
  Interventions: Drug: IZD334; Drug: Placebos

INTERVENTIONS:
Drug: IZD334 — Active Drug
Drug: Placebos — Placebo to Match

SUMMARY:
This is a first in human (FIH), single-centre, double -blind, randomised, cross-over, SAD followed by a MAD study of IZD334 conducted in healthy adult participants as well as an open-label cohort in adult patients with CAPS. The study is designed to evaluate the safety, tolerability, PK, PD, and food effect of IZD334 in healthy adult participants, and to evaluate the safety, tolerability, PK, PD, and preliminary clinical efficacy of IZD334 in adult patients with CAPS.

ELIGIBILITY:
Inclusion Criteria: (Healthy Volunteers)

* Healthy male or female volunteers, aged 18 to 65 years (inclusive at the time of informed consent)
* Participants must be in good general health, with no significant medical history, have no clinically significant abnormalities on physical examination at Screening and/or before administration of the initial dose of study drug
* Participants must have a Body Mass Index (BMI) between ≥18.0 and ≤32.0 kg/m2 at Screening
* Participants must have clinical laboratory values within normal range as specified by the testing laboratory, unless deemed not clinically significant by the Investigator or delegate

Inclusion Criteria: (CAPS Patients)

*Patients with a confirmed diagnosis of CAPS (FCAS or MWS) aged 18 to 65 years (inclusive at the time of informed consent)

Exclusion Criteria: (Healthy volunteer)

* Pregnant or lactating at Screening or planning to become pregnant (self or partner) at any time during the study, including the follow-up period
* Prior or ongoing medical conditions, medical history, physical findings, or laboratory abnormality that, in the Investigator's (or delegate's) opinion, could adversely affect the safety of the participant
* Presence of any underlying physical or psychological medical condition that, in the opinion of the Investigator, would make it unlikely that the participant will comply with the protocol or complete the study per protocol
* Blood donation or significant blood loss within 60 days prior to the first study drug administration

Exclusion Criteria: (CAPS Patients)

* Live vaccinations within 3 months prior to Screening, for the duration of the study and for up to 3 months following the last dose of study drug;
* Positive QuantiFERON test at the Screening visit or within 2 months prior to Screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-09-13 (Actual); Primary Completion 2020-02-04 (Actual); Study Completion 2020-02-04 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events [Safety and Tolerability] | Day 1-8 for SAD
  Incidence, frequency and severity of treatment emergent adverse events.
Incidence of treatment emergent adverse events [Safety and Tolerability] | Day 1-16 for MAD
  Incidence, frequency and severity of treatment emergent adverse events.
Peak plasma concentration (Cmax) single dose | Day 1-3
  Peak plasma concentration following single dose administration
Area under the plasma concentration versus time curve (AUC)- single dose | Day 1-3
  AUC following single dose administration
Peak Plasma Concentration (Cmax)-multiple dose | Days 1-9
  Peak plasma concentration following multiple dose administration
Area under the plasma concentration versus time curve (AUC)- multiple dose | Days 1-9
  AUC following multiple dose administration

SECONDARY OUTCOMES:
Reduction of IL-1 production in stimulated whole blood | Day 1-3 for SAD and Day 1-9 for MAD]
  % reduction in IL-1 production in stimulated whole blood as measured by ELISA
Reduction in CAPS symptom scores | Day 1-15
  Reduction in Physician Assessed CAPS scores based on 8 point questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jason Lickliter, MBBS, PhD, Principal Investigator — Nucleus Network
Locations (1):
- Nucleus Network, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No